CLINICAL TRIAL: NCT02358798
Title: Respiratory Function at Preschool Age of Children Detected of Cystic Fibrosis in Neonatal Period
Acronym: REVOLMUCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9393
Record Dates: First submitted 2015-01-21; First posted 2015-02-09 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Cystic Fibrosis
Keywords: Time evolution of respiratory function; Longitudinal multicenter monitoring of large cohorts; Preschool aged children; Detection of cystic fibrosis in neonatal period
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preschool aged children detected of CF in neonatal period (Experimental): Preschool aged children detected of Cystic Fibrosis in neonatal period
  Interventions: Other: 3 years-assessment of respiratory function

INTERVENTIONS:
Other: 3 years-assessment of respiratory function

SUMMARY:
The widespread neonatal detection of cystic fibrosis in France since 2002 permits to treat children from birth. New treatments used for young children involve to assess efficacy criteria specific to this population. Standard respiratory function criteria for older children and adults is forced expiratory volume/second.

This technique is not suited for preschool aged children (3 to 6 years old) because they are too old to be sedated and too young and immature to be able to make forced expiration technique that are correct, reproducible and prolonged during more than 1 second.

For preschool aged children, in order to assess distal damage and her consequence, the evaluations are: airway resistance by debit interruption technic (Rint), plethysmographic measure of specific resistance (sRaw), functional residual capacity by Helium dilution technique (CRF He), arterial blood gas measurement, pulmonary clearance index.

All these methods have a better success rate and can be used in alternative or with forced spirometry. However, each of them gives only a part of information on airway and lung damage of detected children. It is necessary to combine them for a better information on overall respiratory damage.

In France, each respiratory function test laboratory uses one or any of these methods in addition to flow-volume curve, in function of his practices and his equipment.

So, respiratory function test of preschool aged children is going to diversify more and more to the detriment of an homogeneity of practices between different centers.

A referent population during a longitudinal multicenter monitoring on large cohorts that describe the evolution of pulmonary function, obtained by a standardized methodology is necessary to assess the efficacy of any new treatment. And, with the homogenization of care of children detected of cystic fibrosis in different centers, the description of natural evolution of pulmonary function by a standardized methodology will improve the discriminative power of measure of respiratory function to assess the presence of a worsening in preschool-aged children.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from cystic fibrosis
* Height between 90 et 130cm
* No respiratory exacerbation since 4 weeks
* Benefit from an insurance disease regime

Exclusion Criteria:

* Law-protected patient
* Patient's parent don't understand french language
* Opposition to participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08-19 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Time evolution of functional residual capacity by Helium dilution technique (CRF He) | at each four yearly routine visits

SECONDARY OUTCOMES:
airway resistance by debit interruption technique (Rint) | at each four yearly routine visits
plethysmographic measure of specific resistance (sRaw) | at each four yearly routine visits
arterial blood gas measurement | at each four yearly routine visits
pulmonary clearance index | at each four yearly routine visits
flow-volume curve | at each four yearly routine visits
measurement of organ damage | at each four yearly routine visits
measurement of tobacco exposition | at each four yearly routine visits
measure of administration antibiotics and antiasthmatics treatments | at each four yearly routine visits
  Comparison of the evolution of these parameters to changing those of a historical cohort evaluated before the introduction of neonatal screening.

CONTACTS AND LOCATIONS:
Overall Officials: MATECKI SM Stephan, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital of Montpellier, Arnaud de Villeneuve, Montpellier, France